CLINICAL TRIAL: NCT04069143
Title: An Open-Label Study to Evaluate the Safety, Tolerability, Kinetics, and Repeatability of the Novel Lysophosphatidic Acid Receptor 1 (LPA1) Positron Emission Tomography (PET) Ligand 18F-BMS-986327
Brief Title: A Study to Evaluate the Safety, Tolerability, Kinetics and Repeatability of 18F-BMS-986327
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IM033-002
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Healthy Participants; Idiopathic Pulmonary Fibrosis (IPF)
Keywords: Healthy Participants; Idiopathic Pulmonary Fibrosis (IPF)
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 (Experimental)
  Interventions: Diagnostic Test: 18F-BMS-986327
- Part 2 (Experimental)
  Interventions: Diagnostic Test: 18F-BMS-986327
- Part 3 (Experimental)
  Interventions: Diagnostic Test: 18F-BMS-986327

INTERVENTIONS:
Diagnostic Test: 18F-BMS-986327 — Imaging Agent

SUMMARY:
The purpose of this study is to assess the safety, tolerability, kinetics and test-retest repeatability of the novel LPA1 positron emission tomography (PET) ligand 18F-BMS-986327 in healthy participants and participants with idiopathic pulmonary fibrosis (IPF).

ELIGIBILITY:
Inclusion Criteria:

All Participants:

· Body mass index of 18.0 to 34.0 kg/m^2, inclusive, and body weight ≥ 50 kg

Healthy Participants:

* Male and female healthy volunteers ages 18 or age or older
* No clinically significant deviation from normal in medical history, physical examination, electrocardiograms (ECGs) and clinical laboratory determinations

Idiopathic Pulmonary Fibrosis (IPF) Participants:

* Male and female participants aged 40 to 90 years
* Diagnosis of IPF less than 6 years before randomization
* Have no features supporting an alternative diagnosis on transbronchial biopsy, bronchoalveolar lavage or surgical lung biopsy

Exclusion Criteria (all participants):

* Severe motor problems that prevent the ability to lie still for PET imaging procedure
* Significant acute or chronic medical illness in the opinion of the investigator in consultation with the BMS Medical Monitor, could jeopardize the subject's safety, tolerability, or pharmacokinetics of 18F-BMS-986327
* Current or recent (within 3 months of study drug administration) gastrointestinal disease that could impact upon the absorption of study drug
* Any major surgery within 4 weeks of study drug administration

Other protocol-defined criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 3 days after participant's participation
Incidence of serious adverse events (SAEs) | Up to 30 days after participant's participation
Radiation dosimetry calculated from positron emission tomography-computed tomography (PET-CT) images | 30 days after participant's participation
Test-retest repeatability | 30 days after participant's participation
Biodistribution and lung uptake calculated from PET-CT images in participants with IPF | 30 days after participant's participation

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, New Haven, Connecticut, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm